CLINICAL TRIAL: NCT02654119
Title: A Phase II Study of Adjuvant Therapy Using a Regimen of Cyclophosphamide, Paclitaxel With Trastuzumab in Stage I-II HER2/Neu Positive Breast Cancer Patients
Brief Title: Cyclophosphamide, Paclitaxel, and Trastuzumab in Treating Stage I-II HER2/Neu Positive Breast Cancer After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0318-15-FB; NCI-2015-01879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HER2 Positive Breast Carcinoma; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Paclitaxel; Taxes; Trastuzumab; PF-05280014; Ogivri

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cyclophosphamide, paclitaxel, trastuzumab) (Experimental): SYSTEMIC THERAPY: Patients receive cyclophosphamide IV over 1 hour, paclitaxel IV over 3 hours, and trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE TRASTUZUMAB THERAPY: Beginning in course 6, patients receive trastuzumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Patients may undergo radiation therapy at the discretion of the radiation oncologist and medical oncologist and patients with estrogen/progesterone receptor positive tumors receive hormonal therapy as determined by the medical oncologist per standard NCCN guidelines.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Trastuzumab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014; Trastuzumab-dkst

SUMMARY:
This phase II trial studies the side effects and how well cyclophosphamide, paclitaxel, and trastuzumab work when given after surgery in treating patients with stage I-II human epidermal growth factor receptor (HER2/neu) positive breast cancer (confined to the breast or the breast and lymph nodes under the arm). Drugs used in chemotherapy, such as cyclophosphamide and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as trastuzumab, may interfere with the ability of tumor cells to grow and spread. Giving cyclophosphamide, paclitaxel, and trastuzumab after surgery may help prevent the cancer from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and ability to complete the planned treatment of a dose-dense regimen of cyclophosphamide and paclitaxel with trastuzumab in subjects with newly diagnosed stage I-II HER2/neu positive breast cancer.

II. To estimate recurrence free survival of a dose-dense regimen of cyclophosphamide and paclitaxel with trastuzumab in subjects with newly diagnosed stage I-II HER2/neu positive breast cancer.

OUTLINE:

SYSTEMIC THERAPY: Patients receive cyclophosphamide intravenously (IV) over 1 hour, paclitaxel IV over 3 hours, and trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE TRASTUZUMAB THERAPY: Beginning in course 6, patients receive trastuzumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

Patients may undergo radiation therapy at the discretion of the radiation oncologist and medical oncologist and patients with estrogen/progesterone receptor positive tumors receive hormonal therapy as determined by the medical oncologist per standard National Comprehensive Care Network (NCCN) guidelines.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed stage I-II HER2/neu positive breast cancer
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Within 30 days prior to enrollment: Absolute neutrophil count greater than or equal to 1,500/mcl
* Within 30 days prior to enrollment: Platelet count equal to or greater than 150,000/mcl
* Within 30 days prior to enrollment: Hemoglobin > 11 gm/dl
* Within 30 days prior to enrollment: Alkaline phosphatase equal or less than 1.5 times the upper limit of normal (ULN)
* Within 30 days prior to enrollment: Total bilirubin equal to or less than 1.5 times the ULN
* Within 30 days prior to enrollment: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no greater than 1.5 times the ULN
* Within 30 days prior to enrollment: Creatinine less than 1.5 times the ULN
* Able to give informed consent
* All included subjects must have normal cardiac function as defined by an ejection fraction of > 50% by echocardiogram
* Able to return for treatment and follow-up on the specified days

Exclusion Criteria:

* Prior malignancy; except for adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas
* Subjects with pre-existing grade II peripheral neuropathy
* History of previous chemotherapy
* Stage IV or metastatic breast cancer
* Pregnant or nursing women
* Inability to cooperate with treatment protocol
* No active serious infections or other conditions precluding chemotherapy
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol e.g. unstable angina, myocardial infarction within 6 months, severe infection, etc.
* Known hypersensitivity to any component of required drugs in the study
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C or active hepatitis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiographic (ECG) abnormality at screening has to be documented by the investigator as not medically relevant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of neutropenia, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 | Up to 3 months after final chemotherapy treatment (including trastuzumab)
  The incidence rates of neutropenia and adverse events will be summarized using frequencies, percentages and 90% confidence intervals. Adverse events will be described by cycle. The frequency of toxicity, categorized by toxicity grades, will be summarized.
Incidence of paclitaxel-related neuropathy, graded according to the NCI CTCAE v4.03 | Up to 3 months after final chemotherapy treatment (including trastuzumab)
  The incidence rates of paclitaxel-related neuropathy and adverse events will be summarized using frequencies, percentages and 90% confidence intervals. Adverse events will be described by cycle. The frequency of toxicity, categorized by toxicity grades, will be summarized.
Incidence of grade 3/4 cardiotoxicity, graded according to the NCI CTCAE v4.03 | Up to 3 months after final chemotherapy treatment (including trastuzumab)
  The incidence rates of grade 3/4 cardiotoxicity and adverse events will be summarized using frequencies, percentages and 90% confidence intervals. Adverse events will be described by cycle. The frequency of toxicity, categorized by toxicity grades, will be summarized.
Incidence of grade 3/4 nausea/vomiting, graded according to the NCI CTCAE v4.03 | Up to 3 months after final chemotherapy treatment (including trastuzumab)
  The incidence rates of grade 3/4 nausea/vomiting and adverse events will be summarized using frequencies, percentages and 90% confidence intervals. Adverse events will be described by cycle. The frequency of toxicity, categorized by toxicity grades, will be summarized.
Recurrence free survival (RFS) | First date of therapy until the first notation of clinical progression, relapse or death from any cause, assessed at 2 years
  RFS and survival curves will be plotted following the method of Kaplan and Meier using the full analysis set.
Incidence of inability to complete treatment, defined as a patient that requires a lower dose of therapy (defined as dose lowered by 50%), or a postponement of scheduled treatment of longer than 28 days, or discontinuation of treatment for any reason | Up to 2 years
  Inability to complete treatment will be described using frequencies and proportions and 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Amulya Yellala, MD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska